CLINICAL TRIAL: NCT04896567
Title: Isolation of Cells From Biopsy Tissue to Aid in Kidney Repair
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Superseded by a separate study
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: awaiting IRB approval
Record Dates: First submitted 2018-08-31; First posted 2021-05-21 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Kidney Diseases; Endothelial Dysfunction
MeSH Terms: conditions — Kidney Diseases | interventions — Cell Separation

STUDY DESIGN:
Intervention Model Description: Consecutive patients will be consented to obtain kidney biopsy material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will have kidney biopsy designated for cell isolation and culture.
  Interventions: Diagnostic Test: Cell isolation

INTERVENTIONS:
Diagnostic Test: Cell isolation — Tissue from kidney biopsy will be used to isolate Cluster Differentiation 34+ cells.

SUMMARY:
Endothelial progenitor cells that reside in renal vasculature may be stimulated to initiate differentiation programs during episodes of injury. It is hypothesized that endothelial progenitor cells resident in the kidney can transition to a post-injury phenotype that promotes endothelial repair.

DETAILED DESCRIPTION:
Endothelial dysfunction is central to the pathophysiology of vascular ischemia, bacterial sepsis, toxin-induced thrombotic microangiopathy, and antibody-mediated kidney transplant rejection and often manifest with renal failure. With each of these diagnoses circulating components of the complement cascade bind to endothelial cells and induce disease progression through anaphylactic cellular messaging, monocyte homing, and direct cell membrane disruption. In response to injury during embryologic development avascular metanephric blastema initiate endothelial differentiation. Although circulating hematopoietic progenitor cells have shown therapeutic promise they incorporate into renal vasculature at very low density.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who have a clinical indication for kidney biopsy will be considered.
* All subjects will be at least 18 years of age and may be of any gender.
* Patients undergoing a native or kidney transplant biopsy will be considered.

Exclusion Criteria:

* Patients not undergoing a kidney biopsy will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-21 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cell growth | 1 week
  Tissue will be isolated and cell viability will be documented by rate of colony growth over one week per patient enrolled.

SECONDARY OUTCOMES:
Kidney disease progression | 3 years
  Isolated cell growth will be compared to serum creatinine of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States